CLINICAL TRIAL: NCT05399953
Title: Investigation of Effects of Physioherapy Interventions on Mechanical Properties of Muscle in Head and Neck Cancer
Brief Title: Investigation of Effects of Physiotherapy Interventions on Mechanical Properties of Muscle in Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, FerhatS, PT, MSc, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YeditepeU-Biotechnology
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Cancer; Spinal Accessory Nerve Injury; Thyroid Cancer; Scapular Dyskinesis; Cervical Pain; Shoulder Pain
Keywords: Head and Neck Cancer; Shear Wave Elastography; Myofascial Release; Cancer Rehabilitation; Physiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Accessory Nerve Injuries; Thyroid Neoplasms; Neck Pain; Shoulder Pain | interventions — Myofascial Release Therapy; Exercise

STUDY DESIGN:
Intervention Model Description: A randomized single blind controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Participants in the control group will receive usual care ( standard physical therapy program)
  Interventions: Other: Exercise; Other: Scar Tissue Massage
- Intervention Group (Experimental): Particiapnts in intervevention group will receive both usual care and myofascial release techniques
  Interventions: Other: Myofascial Release Technique; Other: Exercise; Other: Scar Tissue Massage

INTERVENTIONS:
Other: Myofascial Release Technique — Sternocleidomastoid, Upper trapezius, Suboccipital region, Scalenes, Pectoral release, Scapular and hyoid mobilization techniques.
  Duration: 6 weeks, 1 supervised session per week, and the session lasted 30 minutes.
  Arms: Intervention Group
Other: Exercise — Therapeutic exercise: passive and active range of motion, strengthening and postural exercise in order to improve shoulder and cervical mobility, muscle flexibility, strength and endurance, postural control and movement patterns; 2) stretching of pectoral muscles and serratus anterior; 3) scar tissue massage to reduce scar tissue's stiffness.
  Duration of the intervention: 6 weeks (1 supervised session and 2 individual per week). Each exercise will be done 1-3 sets and 5-10 repetitions.The session lasted 30 minutes.
  Exercise diary will be utilized in order to follow the exercise program.
Other: Scar Tissue Massage — Circular, Up and Down, Side to Side technique

SUMMARY:
As the head and neck cancer (HNC) survival rate has increased and therefore, the focus of post-treatments is to improve the quality of patients' life by decreasing the side effects. Treatment of HNC leads to acute and chronic soft tissue damage, and functional loss. However, patients with HNC need having rehabilitation throughout the post-treatment phase so as to improve functional outcomes because of the long term side effects. Chronic shoulder morbidity is one of the complications after surgery due to spinal accesory nerve injury. Moreover, pain, dysphonia, and musculoskeletal impairments are observed in the individuals after the treatments and the patients also have trouble swallowing problems, loss of taste, dry mouth, trismus, nausea, vomiting, and fatigue during and after therapy. Since there is limited research on the usage of manual therapy techniques in HNC patients, this study aims to investigate muscle changes after surgery and the effectiveness of physiotherapy on muscle material behaviour from a biomechanical perspective by using shear wave elastography. In this respect, the hypothesis is:

H0: Physical therapy interventions do not impact mechanical properties of muscle, pain, quality of life, cervical and shoulder functionality in HNC patients after neck dissection.

H1: Physical therapy interventions will improve mechanical properties of muscle, pain, quality of life, cervical and shoulder functionality in HNC patients after neck dissection.

DETAILED DESCRIPTION:
As the HNC survival rate has increased and therefore, the focus of post-treatments is to improve the quality of patients' life by decreasing the side effects. Treatment of HNC leads to acute and chronic soft tissue damage, and functional loss. However, patients with HNC need having rehabilitation throughout the post-treatment phase so as to improve functional outcomes because of the long term side effects. Chronic shoulder morbidity (70% of patients) is one of the common complications after surgery, whereas 84% of survivors complain of their physical appearance due to the remaining head and neck lymphedema (HNL) after radiotherapy. Moreover, pain, dysphonia, and musculoskeletal impairments are observed in the individuals after the treatments and the patients also have trouble swallowing problems, loss of taste, dry mouth, trismus, nausea, vomiting, and fatigue during and after therapy.

Materials might behave in different stress-strain relationships, and it is represented by a stress-strain curve, a basic descriptor of material.Thanks to the stress-strain diagram, differences between materials can be determined such as stiffness, hardness and toughness. Several concepts describe material properties in addition to a stress-strain diagram. For instance, a homogeneous material is one whose properties are not affected by location within the material, anisotropic material is one whose properties are free of direction, and incompressible material retains its volume during deformation. However, the behaviour of soft tissue is anisotropic due to its fibre contents, its constitutive behaviour is nonlinear and incompressible, and it is heterogeneous material owing to its composition, but it can be homogenized under macroscopic analysis. Due to the complexity of soft tissue, its mechanical behaviour is highly affected by density, collagen and elastin's structural arrangement, topographical site, function, and hydrated matrix of proteoglycans. In other words, mechanical properties of soft tissues are related to shape, genetics, age , physical and chemical environmental conditions like strain rate, osmotic pressure and Ph, temperature, which affects skeletal muscle's contractile properties.

It is known that deformable-body changes shape when it is exposed to an external force. In general, several constitutive relations govern the stress and strain relations, for example, plasticity, viscoelasticity, linear elastic, hyperelasticity so on. It is common to use hyperelastic models (i.e. time-independent) so as to determine the association of the stress-strain of soft tissue, even though the biological soft tissues mechanical behaviour is time-dependent . These models are based on the strain energy density which is the energy stored by a system undergoing deformation.

Disuse and immobilization influence muscle fibres harmfully including decreased muscle strength and neural activation of muscle fibre, muscle atrophy, loss of force production and endurance due to decrease in cross-sectional area (CSA). Jones et al., found that immobilization leads to muscle atrophy by decreasing protein synthesis and increasing protein impairment and loss of muscle mass after two weeks of immobilization. Muscle atrophy can exist in the following injury, during an illness such as cancer, sepsis and long term hospitalization. Shortening of myosin and actin filaments alters mechanical properties of muscle because of length-dependent force production. Moreover, the energy production of skeletal muscles is affected during the disuse period by decreasing fat oxidation and enhancing glycolysis, which is a source of muscle energy. Furthermore, muscle composition is impacted due to disuse and inactivity, mainly in type 1 fibre, which maintains postural control. Since radiotherapy and surgery impact negatively on muscle. For instance, after neck dissection, trapezius muscle atrophy seems to be due to SAN injury. It is found that atrophied trapezius muscle's stiffness was significantly lower because of physiological and intrinsic alterations associated with fatty infiltration and atrophy of muscle It is known that physical training affects muscle architecture, such as fibre type distribution, fascicle length, pennation angle and CSA, and force production. Since physical activity contributes to improving the CSA of skeletal muscle, muscle strength and bulk are increased. Moreover, exercise contributes to increased neural activity, contractile tissue and differentiating fibre type. Muscle mechanical properties may change.

Myofascial techniques are one of the manual therapy interventions which focus on treating fascia. It comprises various techniques and interventions such as acupuncture, dry needling, wet needling with pharmaceuticals, and traditional technical approaches such as strain-counter strain, muscle energy technique, positional release, ischemic compression and myofascial release (MFRT). The effectiveness of MFRT has been shown in various trials in different fields. For instance, MFRTs improve outcomes in individuals having shoulder pain, ankle joint restriction, fibromyalgia and lateral epicondylitis. On the other hand, in the cancer field, since MFRTs perform in addition to a standard rehabilitation program, the effect mechanism of MFRT is unclear in cancer . However, it impacts positively on pain, emotions and cancer-related fatigue.

As stated in the surgery part, inflammatory response leads to fibrosis due to increasing edema and healing proteins. This chronic tension that results in abuse, disuse, overuse and anxiety could cause fascial thickening. Within this regard, fascial work is one of the most important parts for treating fibrosis.

As mentioned before, patients with head and neck cancer suffer from the side effects of the treatment. One of the harmful effects of the treatments mostly causes neck and shoulder muscle atrophy, fibrosis and reduction in functionality level. Therefore, it is important to determine changes in mechanical properties of muscles so as to understand effectiveness of physical therapy interventions in HNC patients. To our knowledge, this study will be the first study to directly investigate how neck and shoulder muscles adapt to physical therapy interventions in the scope of material behaviour in HNC patients after neck dissection.

This study will be conducted in Yeditepe University Research Hospital/ Ear Nose and Throat Department.

ELIGIBILITY:
Inclusion Criteria:

* > 18-year-old
* Having modified or functional neck dissection
* 60< Karnofsky Score
* Spinal accesory nerve injury symptoms, such as dropped and winged scapula and decreased shoulder abduction in physical examination.

Exclusion Criteria:

* Metastasis
* Having Radiotherapy- Chemoradiotherapy
* Having severe psychological problem
* Having previous shoulder injury/ scapular dyskinesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Shoulder pain and disability level | Change from baseline at 6 weeks
  Shoulder Pain and Disability Index
Muscle Stiffness | Change from baseline at 6 weeks
  It will be measured by Shear Wave Elastography in relax and contracted state of muscle Muscles: M. Upper Trapezius, M. Sternocleidomastoid
Muscle Thickness | Change from baseline at 6 weeks
  It will be measured by USG B-mode Muscles: M. Upper Trapezius, M. Sternocleidomastoid, M. Masseter /Bilateral
The Quality of Life | Change from baseline at 6 weeks
  The Functional Assessment of Chronic Illness Therapy system of Quality of Life- Head and Neck (FACT H&N Turkish Version)
Shoulder Abduction | Change from baseline at 6 weeks
  Active range of motion will be measured by goniometer for both side
Shoulder Flexion | Change from baseline at 6 weeks
  Active range of motion will be measured by goniometer for both side
Shoulder External Rotation | Change from baseline at 6 weeks
  Active range of motion will be measured by goniometer for both side
Neck Rotation | Change from baseline at 6 weeks
  Active range of motion will be measured by goniometer for both side
Neck Flexion | Change from baseline at 6 weeks
  Active range of motion will be measured by goniometer for both side
Neck Extension | Change from baseline at 6 weeks
  Active range of motion will be measured by goniometer for both side
Neck Lateral Flexion | Change from baseline at 6 weeks
  Active range of motion will be measured by goniometer for both side

CONTACTS AND LOCATIONS:
Overall Officials: Ali F OKYAR, Dr., Study Director — Yeditepe University
Locations (1):
- Yeditepe University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Chen YH, Lin CR, Liang WA, Huang CY. Motor control integrated into muscle strengthening exercises has more effects on scapular muscle activities and joint range of motion before initiation of radiotherapy in oral cancer survivors with neck dissection: A randomized controlled trial. PLoS One. 2020 Aug 6;15(8):e0237133. doi: 10.1371/journal.pone.0237133. eCollection 2020. PMID 32760097
- [Background] Carvalho AP, Vital FM, Soares BG. Exercise interventions for shoulder dysfunction in patients treated for head and neck cancer. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD008693. doi: 10.1002/14651858.CD008693.pub2. PMID 22513964
- [Background] De Groef A, Van Kampen M, Vervloesem N, Dieltjens E, Christiaens MR, Neven P, Vos L, De Vrieze T, Geraerts I, Devoogdt N. Effect of myofascial techniques for treatment of persistent arm pain after breast cancer treatment: randomized controlled trial. Clin Rehabil. 2018 Apr;32(4):451-461. doi: 10.1177/0269215517730863. Epub 2017 Sep 15. PMID 28914087
- [Background] Eickmeyer SM, Walczak CK, Myers KB, Lindstrom DR, Layde P, Campbell BH. Quality of life, shoulder range of motion, and spinal accessory nerve status in 5-year survivors of head and neck cancer. PM R. 2014 Dec;6(12):1073-80. doi: 10.1016/j.pmrj.2014.05.015. Epub 2014 May 28. PMID 24880060
- [Background] Gane EM, Michaleff ZA, Cottrell MA, McPhail SM, Hatton AL, Panizza BJ, O'Leary SP. Prevalence, incidence, and risk factors for shoulder and neck dysfunction after neck dissection: A systematic review. Eur J Surg Oncol. 2017 Jul;43(7):1199-1218. doi: 10.1016/j.ejso.2016.10.026. Epub 2016 Nov 17. PMID 27956321
- [Background] Huang YC, Lee YY, Tso HH, Chen PC, Chen YC, Chien CY, Chung YJ, Leong CP. The Sonography and Physical Findings on Shoulder after Selective Neck Dissection in Patients with Head and Neck Cancer: A Pilot Study. Biomed Res Int. 2019 Jul 22;2019:2528492. doi: 10.1155/2019/2528492. eCollection 2019. PMID 31428629
- [Background] Huang YP, Zheng YP, Leung SF. Quasi-linear viscoelastic properties of fibrotic neck tissues obtained from ultrasound indentation tests in vivo. Clin Biomech (Bristol). 2005 Feb;20(2):145-54. doi: 10.1016/j.clinbiomech.2004.09.012. PMID 15621318
- [Background] Liu KH, Bhatia K, Chu W, He LT, Leung SF, Ahuja AT. Shear Wave Elastography--A New Quantitative Assessment of Post-Irradiation Neck Fibrosis. Ultraschall Med. 2015 Aug;36(4):348-54. doi: 10.1055/s-0034-1366364. Epub 2014 Aug 29. PMID 25171602
- [Background] McGarvey AC, Hoffman GR, Osmotherly PG, Chiarelli PE. Maximizing shoulder function after accessory nerve injury and neck dissection surgery: A multicenter randomized controlled trial. Head Neck. 2015 Jul;37(7):1022-31. doi: 10.1002/hed.23712. Epub 2014 Jul 11. PMID 25042422
- [Background] McNeely ML, Parliament MB, Seikaly H, Jha N, Magee DJ, Haykowsky MJ, Courneya KS. Effect of exercise on upper extremity pain and dysfunction in head and neck cancer survivors: a randomized controlled trial. Cancer. 2008 Jul 1;113(1):214-22. doi: 10.1002/cncr.23536. PMID 18457329
- [Background] McNeely ML, Parliament MB, Seikaly H, Jha N, Magee DJ, Haykowsky MJ, Courneya KS. Predictors of adherence to an exercise program for shoulder pain and dysfunction in head and neck cancer survivors. Support Care Cancer. 2012 Mar;20(3):515-22. doi: 10.1007/s00520-011-1112-1. Epub 2011 Feb 24. PMID 21347523